CLINICAL TRIAL: NCT02214823
Title: Functional Electrical Stimulation Assisted Cycling (eStimCycle):A Novel Intervention to Improve Outcomes in the Critically Ill
Brief Title: eStimCycle: Early Rehabilitation in Critical Care
Acronym: eStimCycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Associate Professor Sue Berney PhD, BPT (Other)
Responsible Party: Sponsor-Investigator, Associate Professor Sue Berney PhD, BPT, Associate Professor, Head of Physiotherapy, Austin Hospital, University of Melbourne
Organization: University of Melbourne (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACTRN12612000528853
Record Dates: First submitted 2014-08-07; First posted 2014-08-12 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Intensive Care Unit Acquired Weakness (ICUAW)
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FES-Cycling (Experimental): Timeframe: Within 72 hours of ICU admission. Program: Standard care physiotherapy AND up to one hour of supine cycling daily using a cycle ergometer (RT300 supine model Restorative Therapies, Ltd or Letto 300.) attached to a six channel stimulator (SAGE) and 2 additional RT50 wireless stimulator channels.
  One leg will undergo cycling alone without the electrodes turned on (sham) and the other leg will undergo cycling and muscle stimulation. Electrodes will be placed on all major lower limb muscles. Intervention will be provided individually and supervised by a physiotherapist in ICU only. Duration /Intensity: Up to 1 hour at least 5 times a week for 28 days or ICU discharge, if 20 sessions have not occurred at this time, intervention will continue until this is achieved. Intensity of muscle stimulation will be delivered at a level able to cause visible muscle contractions, confirmed by palpation.
  A subgroup of 10 individuals will be involved in biomarker analyses.
  Interventions: Device: FES-Cycling; Other: Standard Care
- Standard Care (Active Comparator): Both groups will receive usual medical and nursing care in the ICU and ward. Both groups (control and intervention) will receive standard care physiotherapy including respiratory and rehabilitation with mobilisation activities such as sitting out of bed, marching on the spot, and mobility training.
  A subgroup of 10 individuals will be involved in biomarker analyses. This will involve collection of muscle biopsy, blood and urine analyses at baseline and ICU discharge.
  Interventions: Other: Standard Care

INTERVENTIONS:
Device: FES-Cycling
  Other Names: Cycle ergometer (RT300 supine model Restorative Therapies, Ltd or Letto 300.), six channel SAGE stimulator and two RT50 wireless stimulator channels.
  Arms: FES-Cycling
Other: Standard Care — standard care physiotherapy including respiratory and rehabilitation with mobilisation activities such as sitting out of bed, marching on the spot, and mobility training.

SUMMARY:
Project Summary: Patients who have a length of stay four or more days in ICU and requiring mechanical ventilation assistance to breathe for more than 48 hours will be invited to participate. Participants will be randomised to either receive Functional Electrical Stimulation (eStimCycle) assisted cycling or standard care. As cycling in bed has previously been shown to improve physical function, patients who receive cycling as a treatment will have one leg that cycles and the other leg that cycles with assistance of electrical stimulation as we want to establish the effectiveness of the addition of electrical stimulation of muscle. Muscle bulk, strength and physical function outcome measures will be measured at baseline, weekly in ICU, ICU discharge and hospital discharge. Cognitive function will also be measured at hospital discharge, 6- and 12-month follow-up. A small group of patients in this study will be invited to provide samples of blood, urine and muscle at ICU admission and discharge to try and determine what happens to muscle in patients who are critically ill.

Significance of the Project: This is an important study because the development of ICU-acquired weakness (ICU-AW) can result in long term limitations in physical function. Early treatment to maintain strong muscles during an intensive care stay may help speed up recovery and enhance participation in other rehabilitation treatments and improve functional activities and cognition. These are important objectives for both patients and their families. In addition understanding why the muscles become so weak so quickly in patients in ICU will help to develop treatments that may help to maintain muscle strength.

Study Hypotheses:

Hypothesis 1: eStimCycle versus usual care rehabilitation will improve muscle strength at hospital discharge.

Hypothesis 2: eStimCycle versus usual care rehabilitation will improve cognitive function at 6 month follow up.

Hypothesis 3: Patients receiving eStimCycle will have improved activity of anabolic signalling pathways and less atrophy of skeletal muscle fibre size compared with usual care rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years,
2. expected mechanical ventilation or ECMO >48 h with evidence of systemic inflammation as defined by American College of Chest Physicians (ACCP) Consensus Conference Criteria and
3. predicted ICU length of stay ≥4 days.

Exclusion Criteria:

1. Known primary systemic neuromuscular disease or intracranial process on ICU admission
2. Lower limb amputation/s
3. Unable to perform study physical outcome measures pre morbidly due to condition impairing mobility
4. Assessed by medical staff as not-expected to survive ICU
5. Pregnancy
6. BMI > 40
7. Presence of external fixator or superficial metal in lower limb
8. Open wounds or skin abrasions at electrode application points
9. Presence of cardiac or diaphragmatic pacemaker or implanted defibrillator with no underlying rhythm, as confirmed by the treating physician
10. Transferred from another ICU after > 2 days of mechanical ventilation
11. Platelets < 40 000 and INR > 1.6 (for muscle biopsy)
12. Lower limb malignancy
13. Pre-existing intellectual disability or cognitive impairment limiting the ability to accurately follow instructions.
14. Non-English speaking background restricting the individuals ability to accurately and consistently follow instructions.

Exclusion criteria for the 6 and 12 month cognitive testing follow-up portion of the study:

1. Cognitive impairment (IQCODE >3.3) done by proxy after informed consent obtained
2. No fixed home address
3. Score >= 10 on Alcohol use disorders and identification test (AUDIT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Muscle mass and cross sectional area | Baseline, weekly in ICU for an average 2 weeks and at CU discharge (on average 14 days) with participants beng followed for the duration of hospital stay, an expected average of 4 weeks
  Bioimpedance Spectroscopy will be used to evaluate changes in muscle mass. Ultrasonography of the quadriceps will assess changes in muscle thickness and cross sectional area
Muscle Strength | Baseline, weekly in ICU for an average 2 weeks and at ICU discharge (on average 14 dats) with participants beng followed for the duration of hospital stay on average of 4 weeks. Hand-held dynamometry will also be assessed at 6 and 12 months.
  This will be assessed using the Medical Research Council Scale for identifying muscle weakness in ICU and also hand-held dynamometry for grip strength and isometric quadriceps strength
Neuropsychological Battery of Tests | 6 and 12 months post ICU discharge
  Including the following tests: Hayling Sentence Completion, Weschler Adult Intelligence Scale (Digit Span and Similarities), Weschler Memory III (Logical Memory 1 and 2) and Cognistat (Judgment and Orientation), and Controlled Oral Word Association

SECONDARY OUTCOMES:
Biomarker analyses | Baseline and ICU discharge with an expected average stay of 14 days
  Muscle biopsy, 24 hour urine collection and blood analyses in subgroup of n=20 from main pilot randomised controlled trial.
Hours of mechanical ventilation, ICU hours and ICU readmission | trial completion
  This will be collected from medical records data. This will all be reported at the completion of the trial
Confusion Assessment Method for ICU (CAM-ICU) | Daily in ICU for an expected average of 14 days
  The CAM-ICU is a tool for screening for delirium in critically ill patients.
Montreal Cognitive Assessment (MoCA) | Hospital discharge and expected stay on average of 4 weeks
  A screening tool for cognitive impairment
Activities of Daily Living and Instrumental Activities of Daily Living | Baseline, 90-day status, 6-month call
  Two short and simple questionnaires assessing activities of daily living.
Physical function | Baseline and then weekly until ICU discharge an expected stay on average of 14 days. SPPB and 6MWT will also be measured at hospital discharge with an average length of stay of 4 weeks. 6MWT will be assessed and 6 and 12 months.
  The physical function in ICU test (PFIT), functional status score in the ICU (FSS-ICU), short physical performance battery (SPPB) and six minute walk test (6MWT).
Informant Questionnaire on Cognitive Decline in the Elderly, short form (IQCODE-SF) | Baseline
  The IQCODE-SF for cognitive dysfunction will be completed at baseline by the proxy after obtaining informed consent.
Hospital Anxiety and Depression Scale | 6 and 12 months post recruitment
  A scale used to detect the states of anxiety and depression
Impact of Events Scale - Revised (IES-R) | 6 and 12 months post recruitment
  IES-R is an instrument to measure the subjective response to a specific traumatic event, especially in the response sets of intrusion (intrusive thoughts, nightmares, intrusive feelings and imagery, dissociative-like re-experiencing), avoidance (numbing of responsiveness, avoidance of feelings, situations, and ideas), and hyperarousal (anger, irritability, hypervigilance, difficulty concentrating, heightened startle), as well as a total subjective stress IES-R score.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Denehy, PhD, Principal Investigator — University of Melbourne; Susan Berney, PhD, Principal Investigator — Austin Health; Dale Needham, PhD, Principal Investigator — Johns Hopkins University; Jennifer Paratz, PhD, Principal Investigator — Royal Brisbane and Women's Hospital
Locations (4):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Duke University, Durham, North Carolina
- Australia (2):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Austin Hospital, Melbourne, Victoria

REFERENCES:
- [Background] Parry SM, Berney S, Koopman R, Bryant A, El-Ansary D, Puthucheary Z, Hart N, Warrillow S, Denehy L. Early rehabilitation in critical care (eRiCC): functional electrical stimulation with cycling protocol for a randomised controlled trial. BMJ Open. 2012 Sep 13;2(5):e001891. doi: 10.1136/bmjopen-2012-001891. Print 2012. PMID 22983782
- [Background] Parry SM, Berney S, Granger CL, Koopman R, El-Ansary D, Denehy L. Electrical muscle stimulation in the intensive care setting: a systematic review. Crit Care Med. 2013 Oct;41(10):2406-18. doi: 10.1097/CCM.0b013e3182923642. PMID 23921276
- [Background] Parry SM, Berney S, Warrillow S, El-Ansary D, Bryant AL, Hart N, Puthucheary Z, Koopman R, Denehy L. Functional electrical stimulation with cycling in the critically ill: a pilot case-matched control study. J Crit Care. 2014 Aug;29(4):695.e1-7. doi: 10.1016/j.jcrc.2014.03.017. Epub 2014 Mar 26. PMID 24768534
- [Derived] Berney S, Hopkins RO, Rose JW, Koopman R, Puthucheary Z, Pastva A, Gordon I, Colantuoni E, Parry SM, Needham DM, Denehy L. Functional electrical stimulation in-bed cycle ergometry in mechanically ventilated patients: a multicentre randomised controlled trial. Thorax. 2021 Jul;76(7):656-663. doi: 10.1136/thoraxjnl-2020-215093. Epub 2020 Dec 15. PMID 33323480
- [Derived] Parry SM, Denehy L, Beach LJ, Berney S, Williamson HC, Granger CL. Functional outcomes in ICU - what should we be using? - an observational study. Crit Care. 2015 Mar 29;19(1):127. doi: 10.1186/s13054-015-0829-5. PMID 25888469